CLINICAL TRIAL: NCT06273345
Title: OLIGOS: Impact of Treatment on Primary Tumour in Patients With Newly Diagnosed Oligometastatic Neoplasia of the Prostate
Acronym: OLIGOS
Status: Recruiting | Type: Observational
Sponsor: Istituto Oncologico Veneto IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: IOV-PR-1-2022-OLIGOS
Record Dates: First submitted 2024-02-06; First posted 2024-02-22 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Oligometastatic Prostate Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single arm

SUMMARY:
The proposed study consists of a multicentre prospective observational study involving patients with oligometastatic prostatic neoplasia defined according to CHAARTED criteria.

The aim of the study is the creation of a registry including patients with newly diagnosed OMPCa, belonging to the main urological centres in the Triveneto region, in order to evaluate the oncological outcomes and the impact on the quality of life of local treatment of the primary neoplasm (surgical or radiotherapy) in addition to systemic hormonal treatment (ADT as monotherapy or in combination with Docetaxel/androgen receptor signal inhibitors (ARTA)).

The above criteria define 'high metastatic volume' disease with the following parameters

* ≥ 4 bone metastases, including at least one outside the spine and pelvis
* Presence of visceral metastases Consequently, patients included in the study should not have the above-mentioned characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of new-onset prostate neoplasia (any risk category according to EAU guidelines).
* Histological confirmation of disease by prostate biopsies. Absence of neuroendocrine differentiation
* Low volume of metastatic disease defined according to CHAARTED study criteria (< of 4 bone metastases, absence of visceral metastases)
* Patients without previous treatment of primary malignancy (e.g. previous radical prostatectomy, previous RT)
* Patients treated with systemic therapy (ADT as monotherapy or in combination) for less than 6 months prior to enrolment
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Patients eligible for local treatment of primary malignancy and concomitant systemic therapy
* Signature of informed consent

Exclusion Criteria:

* Inability or unwillingness to give written informed consent
* High volume metastatic disease defined according to CHARTEED criteria
* ECOG performance status > 1
* Patients included in other clinical trials
* Contraindications to hormone/systemic therapy administration
* Previous treatment of primary tumour (RP, RT or other treatment of primary tumour)

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of new-onset oligo-metastatic prostatic neoplasia are included in the study. The definition of oligo-metastatic neoplasm is based on the CHARTEED criteria (less than 4 metastases, absence of visceral metastases).
  All patients should undergo staging by conventional imaging techniques (total body bone scintigraphy, CT abdomen with mdc) or with PET-CT (choline or PSMA) and multiparametric prostate MRI to assess the local extension (clinical stage) of the disease, surgical resectability of the disease and radiotherapy planning.
  In addition, individual cases should be discussed in the multidisciplinary oncology group of the enrolling centre. The choice of treatment type will be based on the decision of the multidisciplinary team and the patient's preferences.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-01-23 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | from the start date of the chosen treatment to the date of the subject's death from any cause, up to 3 years
  Impact of primary tumour treatment in addition to systemic therapy on overall survival (OS) in patients with new-onset oligometastatic prostate neoplasia.

SECONDARY OUTCOMES:
Cancer-specific survival | from the start date of the chosen treatment to the subject's death caused by the malignancy, up to 3 years.
  CSS is defined as the time (quantified in months) from the start date of the chosen treatment and the subject's death caused by the malignancy.
CRPCa development | From the date of randomization up to 3 years
  Serum testosterone levels < 50 ng/dL or 1.7 nmol/L in association with biochemical progression or radiological progression
Radiological progression-free survival | From the treatment start date to radiological progression, up to 3 years
  Definition of radiological progression (r-PFS): time from treatment start date to radiological progression (appearance of two or more new lesions on bone scintigraphy or appearance of visceral lesions).
Quality of life assessment | From admission to discharge, assessed up to 3 years
  Assessment of QoL using the EuroQol 5-dimensional 5-level questionnaire (EQ-5D-5L)19
Quality of life assessment | From admission to discharge, assessed up to 3 years
  Assessment of QoL using the EPIC-26 Short Form questionnaire.
Complications | From admission to discharge, assessed up to 3 years
  Evaluation of complications related to radiotherapy treatment, according to CTCAE v5.0 and surgical treatment, evaluated according to the Clavien Dindo classification

CONTACTS AND LOCATIONS:
Locations (12):
- Italy (12):
  - Ospedale di Bressanone, Brixen, Bolzano
  - Casa di Cura Abano Terme, Abano Terme, Padova
  - Ospedale di Dolo, Dolo, Venezia
  - Ospedale di Bassano Del Grappa, Bassano del Grappa, Vicenza
  - Ospedale dell'Angelo - Mestre, Mestre
  - Istituto Oncologico Veneto IRCCS, Padua
  - Azienda Ospedale Università Padova, Padua
  - Ospedale MAter Salutis - Legnago, Padua
  - Ospedali Riuniti Padova Sud, Padua
  - Azienda Sanitaria Universitaria Giuliano Isontina (ASU GI), Trieste
  - Presidio Ospedaliero Universitario Santa Maria della Misericorida (ASU FC), Udine
  - Azienda Ospedaliera Universitaria Integrata - Verona, Verona

IPD SHARING:
Plan to Share IPD: No